CLINICAL TRIAL: NCT03569631
Title: A Randomized, Double-blind, Placebo-controlled, 2-period Crossover Study of BPN14770 in Adult Males With Fragile X Syndrome
Brief Title: A 2-Period Crossover Study of BPN14770 in Adults Males With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BPN14770-CNS-203
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Fragile X Syndrome; FXS; Fra(X) Syndrome
Keywords: Phosphodiesterase Type 4D; PDE4D; Cognitive Dysfunction; Neurocognitive Disorders; Fragile X Syndrome; Fragile X; FXS; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Cognition Disorders; Enzyme Inhibitors; Nootropic Agents; Developmental Disorder; Autism; Autistic Spectrum Disorder; Genetic Disease; Behavioral Disorder; Learning Disorder
MeSH Terms: conditions — Fragile X Syndrome; Cognitive Dysfunction; Neurocognitive Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Cognition Disorders; Developmental Disabilities; Autistic Disorder; Autism Spectrum Disorder; Genetic Diseases, Inborn; Learning Disabilities | interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPN14770 (Experimental): 25mg BPN14770 capsules, one capsule taken twice daily for 12 weeks
  Interventions: Drug: BPN14770
- Placebo (Placebo Comparator): Matching placebo capsules, one capsule taken twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPN14770 — 25 mg BPN14770 capsules
  Arms: BPN14770
Drug: Placebo — Placebo capsules to mimic 25 mg BPN14770 capsules
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, 2-period crossover study to explore the effects of BPN14770 on cognitive function and behavior in subjects with Fragile X Syndrome. Subjects will receive both active treatment with BPN14770 capsules and matching placebo capsules in the course of the study. One treatment will be administered during each of the 12-week study periods.

DETAILED DESCRIPTION:
A total of 30 subjects will be enrolled. The study consists of a screening period of up to 28 days prior to initial treatment, followed by two double-blind treatment periods, each 12 weeks long. A final follow-up visit or phone contact for safety is planned one week after the conclusion of Period 2.

Eligible subjects will be randomized in a blinded, balanced (1:1) fashion to receive either 25 mg BPN14770 capsules or matching placebo capsules during Period 1, followed by the opposite treatment during Period 2. One capsule will be taken twice daily during both double-blind periods.

Subjects will return to the clinic at the end of Weeks 2, 6, and 12 of each study period. Cognitive and behavioral evaluations will be repeated at Weeks 6 and 12 of each Period. Additionally, patients will be monitored for adverse events via a telephone call at the end of Week 1 of each Period, and one week following completion of Period 2 or following early discontinuation.

During clinic visits, adverse effects will be assessed, and laboratory measures, vital signs, and ECGs will be performed. Suicidality risk will also be evaluated at each clinic visit; if a concern is detected, the subject will be referred for further evaluation and treatment. Cognitive and behavioral assessments will be performed during each clinic visit. Pharmacodynamic measures of CNS function will be obtained to evaluated effects of the drug in the brain. Pharmacokinetic samples will be collected to confirm that study drug is present and to estimate plasma exposure at Week 12 of each Period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male aged 18 to 45 years, inclusive.
2. Subject has Fragile X Syndrome with a molecular genetic confirmation of the full Fragile X Mental Retardation (FMR1) mutation (≥200 CGG repetitions).
3. Current treatment with no more than 3 prescribed psychotropic medications. Anti- epileptic medications are permitted and are not counted as psychotropic medications if they are used for treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications.
4. Permitted concomitant psychotropic medications must be at a stable dose and dosing regimen for at least 2 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
5. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
6. Subjects with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure-free for 3 months preceding Screening, or must be seizure-free for 3 years if not currently receiving anti-epileptics.
7. Behavioral and therapy treatments/interventions must be stable for 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication, and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a school program, due to school vacations, are allowed.
8. Subject must be willing to practice barrier methods of contraception while on study, if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.
9. Subject has a parent, legal authorized guardian or consistent caregiver.
10. Subject and caregiver are able to attend the clinic regularly and reliably.
11. Subject is able to swallow tablets and capsules.
12. For subjects who are not their own legal guardian, subject's parent/legal authorized guardian is able to understand and sign an informed consent form to participate in the study.
13. If subject is his/her own legal guardian, he/she can understand and sign informed consent to participate in the study.
14. If subject is not their own legal guardian, the subject provides assent for participation in the study, if the subject has the cognitive ability to provide assent.

Exclusion Criteria:

1. History of, or current cardiovascular, renal, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cerebrovascular, or other systemic disease that would place the subject at risk or potentially interfere with the interpretation of the safety, tolerability, or efficacy of the study medication. Common diseases such as mild hypertension, well-controlled type 2 diabetes mellitus (hemoglobin A1C [Hgb A1C] <6.5%), etc. are allowed per the investigator's judgment as long as they are stable and controlled by medical therapy that is constant for at least 4 weeks before randomization.
2. Renal impairment, defined as serum creatinine > 1.25 x ULN at screening
3. Hepatic impairment, defined as ALT or AST elevation > 2 x ULN at screening. Note:

   LFTs may be repeated after 1 week to evaluate return to acceptable limits; if LFTs remain elevated, subject is ineligible to participate.
4. Clinically significant abnormalities, in the investigator's judgment, in safety laboratory tests, vital signs, or ECG, as measured during Screening.
5. History of substance abuse within the past year, according to investigator assessment.
6. Significant hearing or visual impairment that may affect the subject's ability to complete the test procedures.
7. Concurrent major psychiatric condition (e.g., Major Depressive Disorder, Schizophrenia or Bipolar Disorder) as diagnosed by the investigator. Subjects with additional diagnosis of Autism Spectrum Disorder or Anxiety Disorder will be allowed.
8. Subject has active diseases that would interfere with participation, such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
9. Subject is planning to commence psychotherapy or cognitive behavior therapy (CBT) during the period of the study or had begun psychotherapy or CBT within 4 weeks prior to Screening.
10. Subject is related to anyone employed by the sponsor, investigator, or study staff.
11. Subject has BMI less than 18 or greater than 36.
12. Subject has participated in another clinical trial within the 30 days preceding Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurney ME, Cogram P, Deacon RM, Rex C, Tranfaglia M. Multiple Behavior Phenotypes of the Fragile-X Syndrome Mouse Model Respond to Chronic Inhibition of Phosphodiesterase-4D (PDE4D). Sci Rep. 2017 Nov 7;7(1):14653. doi: 10.1038/s41598-017-15028-x. PMID 29116166
- [Derived] Berry-Kravis EM, Harnett MD, Reines SA, Reese MA, Ethridge LE, Outterson AH, Michalak C, Furman J, Gurney ME. Inhibition of phosphodiesterase-4D in adults with fragile X syndrome: a randomized, placebo-controlled, phase 2 clinical trial. Nat Med. 2021 May;27(5):862-870. doi: 10.1038/s41591-021-01321-w. Epub 2021 Apr 29. PMID 33927413

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A-B: Participants received 25 mg BPN1470 capsules twice daily in Period 1 followed by matching placebo in Period 2.
- Sequence B-A: Participants received placebo in Period 1 followed by 25 mg BPN1477 capsules twice daily in Period 2.
Period: Period 1 (12 Weeks)
Arm/Group | Sequence A-B | Sequence B-A
Started | 15 | 15
Received At Least 1 Dose of Study Drug | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2 (12 Weeks)
Arm/Group | Sequence A-B | Sequence B-A
Started | 15 | 15
Received At Least 1 Dose of Study Drug | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who were randomized and receive at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A-B | Sequence B-A | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (6.82) | 32.1 (8.00) | 31.6 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 0 | 0 | 0
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A Serious Adverse Event (SAE) was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 24 weeks
Population: Safety Population included all participants who were randomized and received at least one dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- BPN14770: Participants received 25 mg BPN14770 capsules twice daily for 12 weeks either in Period 1 or Period 2.
- Placebo: Participants received placebo to match 25 mg BPN14770 capsules twice daily for 12 weeks either in Period 1 or Period 2.
Arm/Group | BPN14770 | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 11 | 8

2. Secondary Outcome: Change From Baseline in National Institute of Health Toolbox Cognitive Battery Modified for Intellectual Disabilities Crystallized Cognition Composite (NIH-TCB CCC) Score
Description: The NIH-TCB is a battery of extensively validated computer-administered cognitive tests administered on an iPad. The Crystallized Composite score assessment includes Picture Vocabulary and Oral Reading Recognition tests. The NIH toolbox standard score has a mean of 100 and standard deviation (SD) of 15. Higher scores indicate better intellectual abilities.
Time Frame: Baseline to Week 12
Population: Completers population included all randomized participants who completed both periods of treatment with no significant protocol violations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BPN14770 | Placebo
Number analyzed (Participants) | 29 | 30
units on a scale | 0.1 (3.45) | -0.9 (7.18)

3. Secondary Outcome: Change From Baseline Between BPN14770 and Placebo Arm in Visual Analog Scale (VAS) Daily Functioning
Description: The VAS was used to measure the severity of Daily Functioning skills, which is a specific behavioral symptom targeted in this study. Parents or caregivers marked this behavior on a visual line on a score from 0 to 100, with higher scores indicating better quality of life.
Time Frame: Baseline to Week 12
Population: Intent-to-Treat (ITT) population included all randomized participants who received at least one dose of treatment and returned for at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Groups:
- BPN41770: Participants received 25 mg BPN14770 capsules twice daily for 12 weeks either in Period 1 or Period 2.
Arm/Group | BPN41770 | Placebo
Number analyzed (Participants) | 30 | 30
millimeters (mm) | 9.4 (27.91) | 6.8 (22.77)

4. Secondary Outcome: Change From Baseline Between BPN14770 and Placebo Arm in VAS Language
Description: The VAS was used to measure the severity of Language skills, which is a specific behavioral symptom targeted in this study. Parents or caregivers marked this behavior on a visual line on a score from 0 to 100, with higher scores indicating better quality of life.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | BPN41770 | Placebo
Number analyzed (Participants) | 30 | 30
millimeters (mm) | 18.2 (21.47) | 15.4 (22.07)

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 24 weeks
Description: Safety Population included all participants who were randomized and received at least one dose of study drug.
Arm/Group | BPN14770 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BPN14770 (N=30) | Placebo (N=30)
Bursitis infective (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BPN14770 (N=30) | Placebo (N=30)
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03569631/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03569631/SAP_001.pdf